CLINICAL TRIAL: NCT03245710
Title: To Investigate the Efficacy and Mechanism of ZBP Powder Product in the Treatment of Osteopenia in Patients With Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201602096
Record Dates: First submitted 2017-02-24; First posted 2017-08-10 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhibai Dihuang powder (Experimental): Arm: Experimental: Zhibai Dihuang Formula powder Zhibai Dihuang Formula powder: Traditional Chinese medicine formula powder product 5g by mouth, after meal, 3 times in one day for 12 weeks
  Interventions: Dietary Supplement: Zhibai Dihuang powder
- placebos (Placebo Comparator): Arm: placebo Comparator placebos 5g by mouth after meal, 3 times in one day for 12 weeks
  Interventions: Other: Placebos

INTERVENTIONS:
Other: Placebos — starch
  Arms: placebos
Dietary Supplement: Zhibai Dihuang powder — the Traditional Chinese Medicine Formula Powder Product
  Arms: Zhibai Dihuang powder

SUMMARY:
This study investigates the efficacy and mechanism of traditional Chinese medicine formula power product in the treatment of osteopenia in patients with pain. Half of participants will receive Chinese medicine formula power product, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Osteoporosis is a major public health problem, resulting in potentially pain and increasing risk of fracture. Treatment of osteoporosis consists of pharmacotherapy, lifestyle measures, dietary changes, mineral supplementation. Traditional Chinese medicine is a major component of health care in Taiwan and provides one treatment alternative for osteoporosis.

Investigators investigate the efficacy and mechanism of traditional Chinese medicine formula powder product in the treatment of osteopenia patients with pain.This trial is a 12 weeks' randomized, placebo-controlled study. The study was approved by the Wan Fang hospital, and signed informed consent was obtained from each participant. 80 Osteopenia participants with pain were enrolled in this study. There were 80 participants aged 50 years or older included. Before random assignment to treatment, participants were at least moderate pain during 2 weeks as identified by visual analogue scale (VAS) for more than 4. Bone mineral density (BMD) of all participants was -2.5 or below without diabetes, hyperthyroidism, hypoparathyroidism, liver or kidney function disorder, ovariectomy, rheumatoid arthritis, bone cancer, ever used hormone agent within 6 months before assignment to treatment, ever used steroids more than 3 week before assignment to treatment, Primary outcome measures were the change of VAS scale, Oswestry Disability Index and WHOQOL-BREF Taiwan at week 1 and 12. Secondary outcome was the genetic loci associated with a susceptibility to osteoprosis treated by traditional Chinese medicine formula powder product.

Result : To provide evidence of the efficacy and mechanisms of ZBP powder product in the treatment of osteoporosis patients with pain.

ELIGIBILITY:
Inclusion Criteria:

1. aged 50 years or older.
2. VAS score≧4.0 in a week.
3. bone mineral density (BMD) of all participants was -2.5 or below.

Exclusion Criteria:

1. diabetes.
2. thyroidism function disorder.
3. parathyroidism function disorder.
4. liver or kidney function disorder.
5. ovariectomy
6. rheumatoid arthritis.
7. bone cancer.
8. ever used hormone agent within 6 months before assignment to treatment.
9. ever used steroids more than 3 months before assignment to treatment.
10. ever used analgesics, excepted acetaminophen, more than 1 week before assignment to treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2020-05-07 (Estimated); Study Completion 2021-03-07 (Estimated)

PRIMARY OUTCOMES:
Pain on the visual-analogue scales (VAS) for back and legs. | baseline and week 12
  A VAS is a 100-mm-long horizontal line that is anchored by word descriptors at each end (no pain and worst pain possible). The patient selects the point on the line that best represents his or her perception of their pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Yu Huang, MD, Principal Investigator — Taipei Municipal WanFang Hospital
Locations (1):
- WanFangH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No